CLINICAL TRIAL: NCT02797730
Title: Study of Impact of Art Therapy Sessions Given to Family Caregivers of Children With Type 1 Diabetes
Acronym: EDUCARTPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EDUCARTPED
Record Dates: First submitted 2016-05-20; First posted 2016-06-13 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Quality of Life
Keywords: Art Therapy; Caregiver's

ARMS (2):
- art-therapy sessions (Experimental): Caregivers will receive 6 art-therapy sessions
  Interventions: Behavioral: art-therapy sessions
- no art-therapy sessions (No Intervention): Caregivers will not receive 6 art-therapy sessions during the evaluation period

INTERVENTIONS:
Behavioral: art-therapy sessions
  Arms: art-therapy sessions

SUMMARY:
Diagnostic of diabetes in childhood brought modification of family way of life, particularly in child and caregivers lifes.

The education patient programs are in France centered on curative competencies of care.

It is possible that art-therapy improve psycho-social competencies The aim of the study is to evaluate art-therapy sessions on quality of life of caregivers

ELIGIBILITY:
Inclusion Criteria:

* one of the family caregivers of child with diabetes enrolled in patient education programs of 3 hospitals (Hospital of Poitiers, Hospital of Niort and Hospital of La Rochelle)
* who accept the study
* ≥ 18 years
* free, with protection of vulnerable adult
* caregivers of child with who have insurance
* with free, enlightened, signed consent

Exclusion Criteria:

* other research participation
* < 18 years
* host family
* with protection of vulnerable adult
* caregivers of child with who have not insurance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
PedsQL Family Impact score to assess Family Quality of Life | 6 weeks

SECONDARY OUTCOMES:
Anxiety score of caregivers | 6 weeks
self esteem score of caregivers | 6 weeks
quality of life score | 6 weeks
satisfaction score | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - La rochelle, La Rochelle
  - NIORT, Niort
  - POITIERS, Poitiers